CLINICAL TRIAL: NCT00514761
Title: A Phase II, Open, Randomized Study to Assess the Efficacy and Safety of AZD6244 vs Capecitabine (Xeloda) in Patients With Colorectal Cancer Who Have Failed One or Two Prior Chemotherapeutic Regimens.
Brief Title: Phase II Efficacy Study of AZD6244 in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00011
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; AZD6244
MeSH Terms: conditions — Colorectal Neoplasms | interventions — AZD 6244; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Xeloda
  Interventions: Drug: Capecitabine
- 2 (Experimental): AZD6244
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — oral vial
  Other Names: ARRY-142886
  Arms: 2
Drug: Capecitabine — oral tablet
  Other Names: Xeloda
  Arms: 1

SUMMARY:
The purpose of the study is to assess if there is benefit when using AZD6244 in the treatment if metastatic colorectal cancer in comparison with another treatment called capecitabine. This study will also assess how safe and well tolerated AZD6244 is.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer
* require treatment but have failed one or two previous chemotherapeutic regimens that must have included oxaliplatin and/or irinotecan
* have World Health Organisation (WHO) performance status 0-2 and life expectancy > 12 weeks

Exclusion Criteria:

* previous therapy with EGFR inhibitor, MEK inhibitor or capecitabine
* any recent surgery, unhealed surgical incision or severe concomitant condition which makes it undesirable for the patient to participate in the study
* nausea and vomiting, chronic gastrointestinal disease or significant bowel resection that would preclude adequate absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Progression event count | assessed after each visit

SECONDARY OUTCOMES:
safety and tolerability | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Clive Morris, MD, Study Director — AstraZeneca; Gill Pover, MD, Study Director — AstraZeneca; Lance Smith, Study Director — AstraZeneca
Locations (3):
- Brazil (3):
  - Research Site, Goiânia
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1172&filename=CSR-D1532C00011.pdf
- See also: CSR-D1532C00011.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1172&filename=CSR-D1532C00011.pdf